CLINICAL TRIAL: NCT05902572
Title: Outcomes of Differentiated Models of Service Delivery for HIV Treatment at Sentinel Sites in Zambia (Sentinel-Zambia)
Brief Title: DSD Models at Zambia Sentinel Sites (SENTINEL 2)
Acronym: SENTINEL2ZA
Status: Active, not recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Health Economics and Epidemiology Research Office (HE2RO), University of the Witwatersrand (Unknown); Clinton Health Access Initiative Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: H-41512; 2021-Mar-012 (Other: ERES-Converge IRB)
Record Dates: First submitted 2023-06-03; First posted 2023-06-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: HIV; Differentiated service delivery; Zambia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIV treatment survey participants: HIV treatment patients eligible to be enrolled in the patient survey
  Interventions: Other: No intervention
- Provider survey participants: HIV treatment providers eligible to be enrolled in the provider survey
  Interventions: Other: No intervention
- Time and motion observation participants: HIV treatment providers eligible to be enrolled in the time and motion observation study
  Interventions: Other: No intervention
- HIV testing survey participants: Individuals presenting for HIV testing eligible to be enrolled in the HIV testing survey
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational data collection only.

SUMMARY:
To achieve global goals for the treatment of HIV, many countries are piloting and scaling up differentiated service delivery models (DSD). A handful of efforts have been formally described and evaluated in the literature; many others are being implemented formally or informally under routine care, without a research or evaluation goal. For most countries however, the investigators have little evidence on progress and challenges at the facility level-the number of patients actually participating in DSD models, health outcomes and non-health outcomes, effects on service delivery capacity and clinic efficiency and operations, and costs to providers and patients.

Alternative Models of ART Delivery: Optimizing Benefits (AMBIT) is a set of data synthesis, data collection, and data analysis activities aimed at generating information for near- and long-term decision making and creating an approach and platform for ongoing evaluation of differentiated models of HIV treatment delivery. The first AMBIT protocol, "Gathering Records to Evaluate Antiretroviral Treatment" (GREAT, Zambia Ref. No. 2019-Sep-030), collects and analyzes comprehensive patient medical record data, allowing us to assess the effect of DSD models on patients' clinical outcomes and to evaluate uptake of DSD models at scale.

The Sentinel-Zambia study, the second AMBIT protocol, is examining the effect of DSD models on patient and provider satisfaction, service delivery capacity and quality, costs to patients, and other outcomes for which data are not routinely collected in patient-level medical records. The first round of Sentinel-SA was conducted in 2021. The AMBIT 2.0 protocol will allow up to four additional annual rounds of data collection, in 2022-2025. The investigators collected clinic aggregate data, conducted surveys of patients and providers, and observed operations at a selected set of 12 Zambian healthcare facilities and their affiliated DSD models in Round 1. Round 2 (2022) and later rounds will collect the same types of data at 12 facilities in Zambia and will expand the study's research questions to include differentiated models of HIV testing and linkage to care. Results are expected to inform Zambian policy makers and other local and international stakeholders on the actual implications of DSD models for patients, health system operations, and healthcare budgets.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the time and motion study are:

* Patient-facing or patient-supporting service provider at the study site (patient-supporting providers include data clerks, pharmacists, etc.)
* Directly or indirectly involved in the site's implementation of ART and DSD models
* Employed in current role at the study site for at least six months
* Provides written informed consent to participate

Inclusion criteria for provider interviews are:

* Direct or indirect service provider at the study site (indirect providers include supervisors, technical advisors, etc.)
* Directly or indirectly involved in the site's implementation of ART and DSD models
* Employed in current role at the study site for at least six months
* Provides written informed consent to participate.

Inclusion criteria for the patient survey are:

* Living with HIV and on ART for at least six months at the study site
* ≥ 18 years old (18 and older considered adult for research purposes in Zambia)
* Enrolled in a specified model of care (including conventional care) up to the target number of participants for that model and have received at least one medication refill under this model
* Provide written informed consent to participate.

Inclusion criteria for the testing survey are:

* Undergoing HIV testing at the study site or other testing site within the catchment area
* ≥ 18 years old (18 and older considered adult for research purposes in Zambia)
* Provide written informed consent to participate.

Exclusion Criteria:

Exclusion criteria for the time and motion study are:

● None.

Exclusion criteria for provider interviews are:

● None.

Exclusion criteria for the patient survey are:

* Unable to communicate in any of the languages into which the questionnaire has been translated or that is known to the research assistant
* Not physically, mentally, or emotionally able to participate in the study, in the opinion of the investigators or study staff.
* Unwilling to take the time required to complete the questionnaire on the day of consent.

Exclusion criteria for the testing survey are:

* Unable to communicate in any of the languages into which the questionnaire has been translated or that is known to the research assistant
* Not physically, mentally, or emotionally able to participate in the study, in the opinion of the investigators or study staff.
* Unwilling to take the time required to complete the questionnaire on the day of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clients using the Zambian public health system and providers employed by that system.
Sampling Method: Non-Probability Sample
Enrollment: 8280 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient survey participants with HIV viral suppression ≤400 copies/ml at most recent test | 12 months after enrollment
  Viral suppression among ART patients enrolled and not enrolled in differentiated service delivery models

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Rosen, MPA, Principal Investigator — Department of Global Health, BU School of Public Health
Locations (1):
- Clinton Health Access Initiative-Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Data that are collected by the study will be made available after protocol closure. Data that are owned by others (e.g. the National Department of Health) cannot be shared by the authors.
Supporting Information: Study Protocol, ICF
Time Frame: Within one year of protocol closure.

REFERENCES:
- [Result] Ntjikelane V, Phiri B, Kaiser JL, Rosen S, Morgan AJ, Huber A, Mokhele I, Tchereni T, Ngoma S, Lumano-Mulenga P, Pascoe S, Scott N. Effect of differentiated service delivery models for HIV treatment on healthcare providers' job satisfaction and workloads in sub-Saharan Africa: a mixed methods study from Malawi, Zambia, and South Africa. Hum Resour Health. 2025 May 26;23(1):25. doi: 10.1186/s12960-025-00993-6. PMID 40420127
- [Result] Mokhele I, Ntjikelane V, Scott NA, Kaiser JL, Morgan AJ, Huber A, Mokgethi NO, Tchereni TH, Phiri W, Kamanga A, Haimbe PM, Lumano-Mulenga P, Nyirenda RK, Pascoe SJS, Rosen S. Are HIV Treatment Clients Offered a Choice of Differentiated Service Delivery Models? Evidence from Malawi, South Africa, and Zambia. Patient Prefer Adherence. 2025 Jun 25;19:1825-1841. doi: 10.2147/PPA.S494679. eCollection 2025. PMID 40585576
- [Result] Mutanda N, Morgan A, Huber A, Scott N, Mokhele I, Tcherini T, Masina T, Nyirenda R, Kamanga A, Lumano-Mulenga P, Rosen S, Pascoe S. Experiences of Testing Negative or Positive for HIV in Malawi, South Africa, and Zambia: A Cross-Sectional Study. AIDS Behav. 2025 Oct 18. doi: 10.1007/s10461-025-04921-6. Online ahead of print. PMID 41108425
- See also: Project website — https://sites.bu.edu/ambit/